CLINICAL TRIAL: NCT01944930
Title: Laparoscopic Narrow Band Imaging for Detection of Occult Cancer Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Desmond H. Birkett, Chair, Department of General Surgery, Lahey Medical Center, Lahey Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-077
Record Dates: First submitted 2013-05-13; First posted 2013-09-18 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal and Gynecologic Malignancies

ARMS (2):
- Narrow Band Imaging Laparoscopy First (Experimental): Study has single cohort assessed in crossover design. In this arm NBI laparoscopy will be performed first, followed by standard white-light laparoscopy.
  Interventions: Device: Laparoscopic narrow band imaging; Device: Standard white-light laparoscopy
- Standard White-Light Laparoscopy First (Experimental): Study has single cohort assessed in crossover design. In this arm standard white-light laparoscopy will be performed first, followed by NBI laparoscopy.
  Interventions: Device: Laparoscopic narrow band imaging; Device: Standard white-light laparoscopy

INTERVENTIONS:
Device: Laparoscopic narrow band imaging
  Other Names: Olympus Evis Exera II CV-180 video processor; Olympus Evis Exera II CLV-180 light source; Olympus EndoEYE surgical videoscope
Device: Standard white-light laparoscopy
  Other Names: Olympus Evis Exera II CV-180 video processor; Olympus Evis Exera II CLV-180 light source; Olympus EndoEYE surgical videoscope

SUMMARY:
Adult patients evaluated at Lahey Clinic with known or suspected gastrointestinal or gynecologic malignancies and with an indication for diagnostic laparoscopy will be offered participation in the study. The proposed study is a randomized, controlled feasibility trial with crossover design. The study's aim is to evaluate the effectiveness of laparoscopic narrow band imaging (NBI) compared to standard white-light laparoscopy for detection of peritoneal cancer metastases. Study patients will undergo laparoscopic evaluation of the peritoneal cavity using a routine white-light videolaparoscope with the capability of NBI. The order of white-light and NBI laparoscopy will be randomized for each patient (crossover design). Frozen-section histopathology biopsies will be retrieved of all suspicious-appearing abnormalities using best clinical practices. The number of detected peritoneal metastases will be compared between each diagnostic laparoscopy technique. To gauge the rate of potentially missed metastases, peritoneal cancer recurrence will be surveyed through a 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diagnosis or suspicion of malignancy of the gastrointestinal or gynecologic tract

Exclusion Criteria:

* clinical contraindication to diagnostic laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schnelldorfer, MD, Study Director — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States

REFERENCES:
- [Derived] Schnelldorfer T, Jenkins RL, Birkett DH, Wright VJ, Price LL, Georgakoudi I. Laparoscopic narrow band imaging for detection of occult cancer metastases: a randomized feasibility trial. Surg Endosc. 2016 Apr;30(4):1656-61. doi: 10.1007/s00464-015-4401-9. Epub 2015 Jul 21. PMID 26194251

RESULTS

PARTICIPANT FLOW:
Groups:
- Narrow Band Imaging Laparoscopy First: Study has single cohort assessed in crossover design. In this arm NBI laparoscopy will be performed first, followed by standard white-light laparoscopy.
  Laparoscopic narrow band imaging
  Standard white-light laparoscopy
- Standard White-Light Laparoscopy First: Study has single cohort assessed in crossover design. In this arm standard white-light laparoscopy will be performed first, followed by NBI laparoscopy.
  Laparoscopic narrow band imaging
  Standard white-light laparoscopy
Period: Overall Study
Arm/Group | Narrow Band Imaging Laparoscopy First | Standard White-Light Laparoscopy First
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrow Band Imaging Laparoscopy First | Standard White-Light Laparoscopy First | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 56 (13) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Detectable Peritoneal Metastases
Description: number of additionally visualized peritoneal lesions
Time Frame: After each Laparoscopy, at time of procedure
Measure: Number; unit: percentage of lesions
Groups:
- Narrow Band Imaging Laparoscopy: Study has single cohort assessed in crossover design. In this arm NBI laparoscopy will be performed first, followed by standard white-light laparoscopy.
  Laparoscopic narrow band imaging
- Standard White-Light Laparoscopy: Study has single cohort assessed in crossover design. In this arm standard white-light laparoscopy will be performed first, followed by NBI laparoscopy.
  Standard white-light laparoscopy
Arm/Group | Narrow Band Imaging Laparoscopy | Standard White-Light Laparoscopy
Number analyzed (Participants) | 20 | 20
percentage of lesions | 0 | 2

ADVERSE EVENTS:
Groups:
- Narrow Band Imaging Laparoscopy First: Study has single cohort assessed in crossover design. In this arm NBI laparoscopy will be performed first, followed by standard white-light laparoscopy. Therefore any adverse event cannot be traced back to each single intervention and can only be described cumulative.
  Laparoscopic narrow band imaging
  Standard white-light laparoscopy
- Standard White-Light Laparoscopy First: Study has single cohort assessed in crossover design. In this arm standard white-light laparoscopy will be performed first, followed by NBI laparoscopy. Therefore any adverse event cannot be traced back to each single intervention and can only be described cumulative.
  Laparoscopic narrow band imaging
  Standard white-light laparoscopy
Arm/Group | Narrow Band Imaging Laparoscopy First | Standard White-Light Laparoscopy First
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No